CLINICAL TRIAL: NCT07269158
Title: A Phase IIb Randomized Clinical Trial of Immune Checkpoint Inhibitor-based Maintenance Therapy in Patients With Advanced Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-1249
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Biliary Tract Neoplasms; Advanced Cancer; Immunotherapy
Keywords: Biliary Tract Neoplasms [including Intrahepatic Cholangiocarcinoma, Extrahepatic Cholangiocarcinoma, and Gallbladder Neoplasms]
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — durvalumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immunotherapy Maintenance (Experimental): Durvalumab or Pembrolizumab
  Interventions: Drug: Durvalumab or Pembrolizumab
- Immunotherapy Maintenance + Lenvatinib (Active Comparator): Durvalumab or Pembrolizumab + Levnatinib
  Interventions: Drug: Durvalumab or Pembrolizumab + Levnatinib
- Immunotherapy Maintenance + Venadaparib (Active Comparator): Durvalumab or Pembrolizumab + Venadaparib
  Interventions: Drug: Durvalumab or Pembrolizumab + Venadaparib
- Immunotherapy Maintenance + SCL-3010 (Active Comparator): Durvalumab or Pembrolizumab + SCL-3010
  Interventions: Drug: Durvalumab or Pembrolizumab + SCL-3010

INTERVENTIONS:
Drug: Durvalumab or Pembrolizumab — Phase 2 Durvalumab 1500mg IV D1, q 4weeks or Pembrolizumab 200mg IV D1, q 3weeks
  Arms: Immunotherapy Maintenance
Drug: Durvalumab or Pembrolizumab + Levnatinib — Durvalumab 1500mg IV D1, q 4weeks or Pembrolizumab 200mg IV D1, q 3weeks Lenvatinib 12mg (≥60 kg) PO q 1cycle or 8mg (<60 kg) PO q 1cycle
  Arms: Immunotherapy Maintenance + Lenvatinib
Drug: Durvalumab or Pembrolizumab + Venadaparib — Durvalumab or Pembrolizumab + Venadaparib
  Arms: Immunotherapy Maintenance + Venadaparib
Drug: Durvalumab or Pembrolizumab + SCL-3010 — Durvalumab or Pembrolizumab + SCL-3010
  Arms: Immunotherapy Maintenance + SCL-3010

SUMMARY:
"Biliary tract cancer (BTC) is a rare malignancy with a poor prognosis. Most patients present with unresectable disease, and even after curative-intent resection, recurrence is common. Since the ABC-02 trial, gemcitabine plus cisplatin (Gem/Cis) has been established as the standard first-line regimen, but the median overall survival (OS) remains approximately 11.7 months. Recent studies combining immune checkpoint inhibitors (ICIs) such as durvalumab or pembrolizumab with Gem/Cis have improved OS to 12.7-12.9 months, establishing ICI-based combination therapy as the new standard. However, the optimal maintenance therapy following initial chemoimmunotherapy remains undefined.

This phase IIb study enrolls patients with advanced BTC who achieved disease control after at least eight cycles of Gem/Cis plus ICI. The trial compares the efficacy and safety of ICI monotherapy maintenance versus ICI in combination with lenvatinib, venadaparib, or interleukin-2 (IL-2, SLC-3010).

Lenvatinib, through inhibition of FGFR2 and modulation of the tumor immune microenvironment, is expected to enhance ICI efficacy. PARP inhibitors may be beneficial in patients with homologous recombination deficiency (HRD) or platinum-sensitive disease. Additionally, IL-2 can activate tumor-infiltrating lymphocytes and alleviate the immunosuppressive microenvironment, potentially augmenting ICI responsiveness.

This study aims to explore a novel maintenance strategy integrating molecular targeted therapy, DNA damage repair modulation, and cytokine-based immunotherapy to overcome the limitations of current ICI monotherapy in BTC. The combination approach is expected to improve disease control and survival outcomes in patients with advanced BTC.

DETAILED DESCRIPTION:
This phase IIb randomized trial assesses the efficacy and safety of immune checkpoint inhibitor (ICI) monotherapy versus ICI-based combination maintenance therapy with lenvatinib, venadaparib, or SLC-3010 in advanced biliary tract cancer. Durvalumab (q4w) or pembrolizumab (q3w) serve as backbone ICIs. For each group, Lenvatinib is given orally once daily, venadaparib orally, or SLC-3010 as a 60-minute IV infusion. Recommended phase II doses will be established via a 3+3 dose-escalation design, with toxicity management per NCI-CTCAE v5.0.

ELIGIBILITY:
Inclusion Criteria:

-Patients with advanced biliary tract cancer who have completed at least 8 cycles of Durvalumab plus Gemcitabine and Cisplatin treatment without radiologic evidence of disease progression, and are planned to receive Durvalumab maintenance therapy.

(Patients treated with Pembrolizumab plus Gemcitabine/Cisplatin are also eligible if they are to continue Pembrolizumab monotherapy without Gemcitabine as maintenance therapy.)

* Patients who are 20 years of age or older at the time of signing the informed consent form.
* Patients with histologically confirmed biliary tract cancer, including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, or gallbladder carcinoma.

(Patients with neuroendocrine tumors or sarcomas are excluded.)

* Patients who are willing and able to provide written informed consent for participation in the study.
* Patients with measurable disease according to RECIST version 1.1.
* ECOG performance status of 0 or 1.
* Estimated life expectancy ≥ 3 months.
* Patients with adequate organ and bone marrow function, without transfusion or administration of hematopoietic growth factors (e.g., G-CSF) within 2 weeks prior to treatment initiation, defined as follows:
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L
* Platelet count ≥ 75 × 10⁹/L
* Serum creatinine ≤ 1.5 × upper limit of normal (ULN), or estimated creatinine clearance ≥ 45 mL/min (calculated using the Cockcroft-Gault formula; see Appendix 7)
* AST and ALT ≤ 3.0 × ULN (≤ 5.0 × ULN if liver metastases are present)
* Total bilirubin ≤ 2.0 × ULN (≤ 3.0 × ULN for patients with Gilbert's syndrome)
* International normalized ratio (INR) ≤ 1.5 or prothrombin time ≤ 1.5 × ULN
* Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
* Women of childbearing potential must agree to use highly effective contraception during the entire study period and for at least 6 months after the last dose of investigational product, and must have a negative serum pregnancy test within 14 days prior to first dose.
* Male patients who have not undergone sterilization must agree to use highly effective contraception during the entire study period and for at least 120 days after the last dose of investigational product.
* Patients who are willing to provide tumor tissue samples obtained by endoscopic biopsy or excisional biopsy.
* Patients who are able to understand and comply with the study procedures and are considered likely to complete the study by the investigator.

Exclusion Criteria:

1. Patients who have received more than 10 cycles of immune checkpoint inhibitor (ICI) plus Gemcitabine and Cisplatin combination therapy for advanced biliary tract cancer.
2. Patients who have been treated for, or have evidence of recurrence or progression of, any malignancy other than biliary tract cancer within the past 3 years.

   Exceptions: Patients who have been disease-free for ≥3 years after curative treatment, or patients with the following malignancies are not excluded: basal cell carcinoma of the skin, Stage I squamous cell carcinoma of the skin, carcinoma in situ, intramucosal carcinoma, or superficial bladder carcinoma.
3. Patients with residual adverse events from prior therapy or surgery that may interfere with the safety evaluation of the investigational product.
4. Patients with a history of hypersensitivity to any component of monoclonal antibody products.
5. Patients with a history or evidence of active, non-infectious interstitial lung disease (pneumonitis).
6. Patients with symptomatic or clinically active brain or leptomeningeal metastases requiring treatment.

   (Patients with asymptomatic, stable, and untreated brain metastases may be enrolled.)
7. Patients who are immunodeficient or are receiving systemic corticosteroids or other immunosuppressive therapy within 7 days prior to the first dose of the investigational product.

   (Physiologic doses of corticosteroids, such as for acute asthma exacerbation, may be allowed after consultation with the principal investigator.)
8. Patients with uncontrolled or significant cardiovascular disease, defined as any of the following:

   * Myocardial infarction within 180 days prior to randomization
   * Uncontrolled angina within 180 days prior to randomization
   * Congestive heart failure classified as New York Heart Association (NYHA) Class III or IV
   * Uncontrolled hypertension despite appropriate therapy (systolic ≥150 mmHg or diastolic ≥90 mmHg for >24 hours)
   * Clinically significant arrhythmia requiring treatment
9. Patients with severe chronic infections or active infections, including active or previously known tuberculosis.
10. Patients with active autoimmune disease that has required systemic treatment (e.g., disease-modifying agents, corticosteroids, or immunosuppressants) within the past 2 years.

    (Replacement therapy, such as thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency, is not considered systemic treatment.)
11. Patients who have received any anticancer therapy other than immune checkpoint inhibitor + Gemcitabine + Cisplatin combination therapy for biliary tract cancer.

    (Adjuvant chemotherapy completed ≥6 months before study drug initiation is permitted.)
12. Patients who have undergone major surgery under general anesthesia within 28 days or minor/local surgery within 14 days before the start of study treatment.

    (Diagnostic procedures such as laparoscopic biopsy may be allowed upon investigator's discretion.)
13. Patients who, in the opinion of the investigator, have any condition, treatment, active or ongoing symptomatic infection, or abnormal laboratory finding that could confound study results, interfere with study participation, or pose undue risk to the patient.
14. Patients with a known history of psychiatric disorders or substance abuse that may interfere with compliance to study requirements.
15. Patients with a known history of human immunodeficiency virus (HIV-1/2) infection.
16. Patients with active hepatitis B (HBsAg-positive and HBV DNA detected) or active hepatitis C (anti-HCV positive with detectable HCV RNA).

    Exception: Patients with inactive or asymptomatic HBV carriers, chronic HBV infection, or non-active HCV infection are eligible if HBV DNA < 500 IU/mL (or < 2500 copies/mL) at screening.
17. Pregnant or breastfeeding women.
18. Patients who have received any unapproved or investigational drug, combination product, or formulation within 28 days prior to the start of study treatment.
19. Any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in this clinical study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase II Dose | Up to 4 years
  Recommended Phase II Dose decided during DLT periods
Phase II: Progression Free Survival(PFS) | Up to 4 years
  Progression-free survival (PFS) is the length of time from the start of treatment until the disease progresses or the patient dies from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate, ORR | Up to 4 years
  Objective response rate (ORR) is the proportion of patients achieving complete response (CR) or partial response (PR) per RECIST 1.1.
Overall Survival, OS | Up to 4 years
  Overall survival (OS) is defined as the time interval from cycle 1 day 1 to death from any cause or last follow-up.
Disease Control Rate, DCR | Up to 4 years
  Disease control rate (DCR) is the proportion of patients with CR, PR, or stable disease (SD) per RECIST 1.1.
Duration of Response, DOR | Up to 4 years
  Duration of response (DOR) is defined as the time interval from the first documented response (CR or PR) per RECIST 1.1 to tumor progression, death, or last follow-up.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 4 years
  Safety per NCI CTCAE v5.0 (Number of participants with treatment-related adverse events as assessed by CTCAE v5.0)
Quality of life (QoL) determined by EORTC QLQ-C30 | Up to 4 years
  QoL determined by EORTC QLQ-C30
Quality of life (QoL) | Up to 4 years
  QoL determined by EORTC QLQ-BIL21.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Medical Oncology, Yonsei Cancer Center, Yonsei Univ. College of Medicine, Korea, Seoul, South Korea